CLINICAL TRIAL: NCT03843099
Title: Decisions About Exercise During Weight Loss: Pilot Study
Brief Title: Physical Activity Choices Everyday- A Pilot Study
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University at Buffalo (Other); Kent State University (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, Amy Gorin, Principal Investigator, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H19-008
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Weight Loss + Healthy Thinking (Active Comparator): Participants will receive a 4-week behavioral weight loss intervention based on evidence-based weight loss strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will be asked to read short passages related to nutrition and a healthy lifestyle through our study website twice a day for the duration of treatment.
  Interventions: Behavioral: Behavioral Weight Loss + Healthy Thinking
- Behavioral Weight Loss + Future Thinking (Experimental): Participants will receive a 4-week behavioral weight loss intervention based on evidence-based weight loss strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will create descriptions of upcoming positive events and will be asked to read short passages through our study website at least twice a day for the duration of treatment.
  Interventions: Behavioral: Behavioral Weight Loss + Future Thinking

INTERVENTIONS:
Behavioral: Behavioral Weight Loss + Future Thinking — Participants will receive a 4-week behavioral weight loss intervention based on evidence-based weight loss strategies focused on diet, exercise, and behavioral skills.
  Arms: Behavioral Weight Loss + Future Thinking
Behavioral: Behavioral Weight Loss + Healthy Thinking — Participants will receive a 4-week behavioral weight loss intervention based on evidence-based weight loss strategies focused on diet, exercise, and behavioral skills.
  Arms: Behavioral Weight Loss + Healthy Thinking

SUMMARY:
This study aims to test two strategies for weight loss. Participants will be randomly assigned to one of the two 4-week weight loss programs: (1) a behavioral weight loss program that involves recording weekly weight, physical activity, and caloric intake plus daily exercises in which information about a healthy lifestyle is reviewed or (2) a behavioral weight loss program that involves recording weekly weight, physical activity, and caloric intake plus daily exercises in which descriptions of positive future events are reviewed. Throughout the study, participants will complete assessments that examine the effects of the interventions on delay discounting, physical activity, weight, and other important health and psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70
* Body Mass Index between 30-50
* English Speaking
* Have a smartphone that can be used for study activities

Exclusion Criteria:

* Report being unable to walk 2 blocks without stopping
* Are currently participating in weight loss treatment, have a history of bariatric surgery, or lost ≥5% in the past 6-months
* Are pregnant or plan to become pregnant within 2 months
* Report a heart condition, chest pain during periods of rest or activity, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Report a medical condition that could jeopardize their safety in a weight control program with diet and exercise guidelines
* History of or current traumatic brain injury, dementia or Alzheimer's disease; a history of Multiple Sclerosis, or other neurological disorders
* Report conditions that, in the judgment of the PI, would render them unlikely to follow the protocol (e.g., relocation, dementia, unable to read and write in English)
* Have no Internet access or unwilling to use personal smartphone for study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Physical Activity | baseline and week 7
  Change in minutes of moderate to vigorous physical activity measured via a waist worn accelerometer during 7 day time periods.
Delay Discounting | baseline and week 7
  Change in delay discounting measured using a choice task.

SECONDARY OUTCOMES:
Weight | 4 weeks
  Weight change from baseline to post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UConn Weight Management Research Laboratory, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No